CLINICAL TRIAL: NCT04166565
Title: Daratumumab Combined With Bortezomib, Cyclophosphamide and Dexamethasone for the Treatment of Multiple Myeloma Patients Presenting With Extramedullary Disease. The ANTARES Study
Brief Title: Daratumumab Combined With Bortezomib, Cyclophosphamide and Dexamethasone for the Treatment of Multiple Myeloma Patients Presenting With Extramedullary Disease
Acronym: EMN19
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Stichting European Myeloma Network (Network)
Collaborators: Janssen, LP (Industry)
Responsible Party: Sponsor
Organization: European Myeloma Network B.V. (Network)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EMN19; 2019-000991-41 (EudraCT Number)
Record Dates: First submitted 2019-11-12; First posted 2019-11-18 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Multiple Myeloma; Extramedullary Plasmacytoma
MeSH Terms: conditions — Multiple Myeloma | interventions — daratumumab; Bortezomib; Cyclophosphamide; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Daratumumab/bortezomib/cyclophospamide/dexamethasone (daraVCD) (Experimental): Daratumumab 16 mg/kg will be administered by i.v. infusion. Daratumumab will be administered weekly in Cycles 1 and 2, then every 2 weeks for Cycles 3-6, and thereafter every month up to 36 months.
  Bortezomib 1.5 mg/m2 bortezomib will be administered by a subcutaneous injection once weekly (Days 1, 8, 15 and 22) in all cycles.
  Cyclophosphamide 300 mg/m2 will be administered as a p.o. or i.v. weekly dose (Days 1, 8, 15, and 22) in every 28-day cycle (maximum weekly dose 500 mg).
  Dexamethasone will be administered on Days 1, 2, 8, 9, 15, 16, 22 and 23 in all cycles. On daratumumab infusion days dexamethasone may be administered i.v. or p.o. approximately 1 hour before the daratumumab infusion. On days when daratumumab is not administered, dexamethasone is to be administered p.o.
  Interventions: Drug: Daratumumab; Drug: Bortezomib; Drug: Cyclophosphamide; Drug: Dexamethasone

INTERVENTIONS:
Drug: Daratumumab — Daratumumab 16 mg/kg will be administered by i.v. infusion. Daratumumab will be administered weekly in Cycles 1 and 2, then every 2 weeks for Cycles 3-6, and thereafter every month up to 36 months.
Drug: Bortezomib — Bortezomib 1.5 mg/m2 bortezomib will be administered by a subcutaneous injection once weekly (Days 1, 8, 15 and 22) in all cycles.
  Other Names: Velcade
Drug: Cyclophosphamide — Cyclophosphamide 300 mg/m2 will be administered as a p.o. or i.v. weekly dose (Days 1, 8, 15, and 22) in every 28-day cycle (maximum weekly dose 500 mg).
  Dexamethasone will be administered on Days 1, 2, 8, 9, 15, 16, 22 and 23 in all cycles. On daratumumab infusion days dexamethasone may be administered i.v. or p.o. approximately 1 hour before the daratumumab infusion. On days when daratumumab is not administered, dexamethasone is to be administered p.o.
Drug: Dexamethasone — Dexamethasone will be administered on Days 1, 2, 8, 9, 15, 16, 22 and 23 in all cycles. On daratumumab infusion days dexamethasone may be administered i.v. or p.o. approximately 1 hour before the daratumumab infusion. On days when daratumumab is not administered, dexamethasone is to be administered p.o.

SUMMARY:
This trial will try to establish the feasibility and efficacy of the combination of DaraVCD in Multiple Myeloma (MM) patients presenting with extramedullary disease (EMD). The study will be conducted as a Phase II trial.

Forty patients will be included in the study cohort. All patients will be followed closely for toxicities and response assessment. After completion of treatment, patients will be followed every 6 months for survival until 5 years after enrolment

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed diagnosis of Multiple Myeloma(MM) (IMWG consensus guidelines)
2. Newly diagnosed or relapsed (patients should have received a maximum of one line of prior therapy) patients presenting with extramedullary disease (EMD) of the skin, liver, lungs, central nervous system, lymph nodes or other tissues, but not solely paraskeletal plasmacytoma (expanding soft tissue masses)* detected by physical exam and confirmed (when required) by Weight Bearing CT/MRI/PET-CT and/or biopsy**. Documentation of plasma cell infiltration is highly recommended unless it requires invasive surgical intervention such as intracerebral infiltration of plasmacytomas.

   *Note: patients with only paraosseous extension of MM forming soft tissue plasmacytomas are not eligible

   **Note: An additional radiologic assessment at screening is not required to confirm EMD. Documentation in terms of physician's/pathologist's report and/or radiologic assessments performed within 42 days of C1D1 will suffice for the purposes of eligibility. All patients however will undergo a baseline radiologic assessment at C1D1 for response purposes.
3. Patients with one prior line of therapy must have:

   * achieved a response (PR or better based on investigator's determination of response by the IMWG criteria) to at least one prior regimen.
   * documented evidence of PD based on Investigator's determination of response as defined by the IMWG criteria on or after the last line of treatment.
4. Age ≥ 18 years
5. Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2. Note: for patients with central nervous system (CNS) involvement, an ECOG performance status >2 is also acceptable
6. Each patient must sign an informed consent form (ICF) indicating that he or she understands the purpose of and procedures required for the study and are willing to participate in the study. Patients must be willing and able to adhere to the prohibitions and restrictions specified in this protocol, as referenced in the ICF.
7. Patient must have measurable disease of MM as defined by the below criteria:

   * IgG MM: Serum M protein level ≥1.0 g/dL or urine M protein level ≥200 mg/24 hours, or
   * IgA, IgD, IgE, IgM MM: Serum M-protein level ≥0.5 g/dL or urine M-protein level ≥200 mg/24 hours; or
   * Light chain MM, for patients without measurable disease in the serum or urine: Serum immunoglobulin free light chain (FLC) ≥10 mg/dL and abnormal serum immunoglobulin kappa lambda FLC ratio.
8. Reproductive Status

   * Women of childbearing potential (WOCBP) must have a negative serum or urine pregnancy test at screening. Females are not of childbearing potential if they have been in natural menopause for at least 24 consecutive months, or have had a hysterectomy and/or bilateral oophorectomy
   * Women must not be breastfeeding
   * WOCBP must agree to follow instructions for reliable methods of birth control. This includes one highly effective (< 1% failure rate per year) form of contraception (tubal ligation, intrauterine device (IUD), combined or progestogen only hormonal contraception associated with inhibition of ovulation [birth control pills, injections, hormonal patches, vaginal rings or implants] or partner's vasectomy) and one additional effective contraceptive method (male latex or synthetic condom, diaphragm, or cervical cap). Contraception must begin 4 weeks before the start of treatment and continue for the duration of study treatment and for 3 months after cessation of daratumumab or 12 months after cessation of cyclophosphamide, whichever is longer.
   * Males who are sexually active must always use a latex or synthetic condom during any sexual contact with females of reproductive potential, even if they have undergone a successful vasectomy. They must also agree to follow instructions for methods of contraception for 4 weeks before the start of study treatment, for the duration of study treatment, and for 3 months after cessation of daratumumab or 6 months after cessation of cyclophosphamide, whichever is longer.
   * Female patients must not donate eggs for up to 3 months after cessation of daratumumab or 12 months after cessation of cyclophosphamide, whichever is longer.
   * Male patients must not donate sperm for up to 3 months after cessation of daratumumab or 6 months after cessation of cyclophosphamide, whichever is longer.
   * Azoospermic males and WOCBP who are not heterosexually active are exempt from contraceptive requirements. However, WOCBP will still undergo pregnancy testing as described above.

Exclusion Criteria:

1. Solitary plasmacytoma
2. Paraosseous extension of MM forming soft tissue plasmacytomas only (without EMD).
3. Previous therapy with any anti-CD38 or anti-CS1 monoclonal antibody
4. Patients refractory to bortezomib based regimens (PD on or within 60 days of completion of bortezomib OR failure to achieve at least a minimal response [MR]) as the prior line of therapy
5. Patients who have Bortezomib or Daratumumab hypersensitivity
6. Patients who have active or chronic infections
7. Patients who have received anti-myeloma treatment within 2 weeks or 5 pharmacokinetic half-lives of the treatment, whichever is longer, before Cycle 1 Day 1 (C1D1). The only exception is emergency use of a short course of corticosteroids (equivalent of dexamethasone 40 mg/day for a maximum of 4 days) for palliative treatment before C1D1.
8. Previous autologous stem cell transplant (ASCT) within 12 weeks before C1D1.
9. Previous allogenic stem cell transplant (alloSCT) regardless of timing.
10. Patient has received radiotherapy within 14 days from C1D1. NOTE: Urgent localized radiotherapy for Spinal Cord Compression or Central Nervous System Involvement is allowed.
11. Patient has known chronic obstructive pulmonary disease (COPD) with a Forced Expiratory Volume in 1 second (FEV1) <50% of predicted normal. Note that FEV1 testing is required for patients suspected of having COPD and patients must be excluded if FEV1 <50% of predicted normal
12. Patient has known moderate or severe persistent asthma within the past 2 years (see) or currently has uncontrolled asthma of any classification. Note: Patients who currently have controlled intermittent asthma or controlled mild persistent asthma are allowed in the study).
13. Severe cardiovascular disease (arrhythmias [CTCAE Grade 3 or higher] requiring chronic treatment, congestive heart failure [New York Heart Association (NYHA) Class III - IV] or symptomatic ischemic heart disease);
14. Severe pulmonary dysfunction (CTCAE grade 3-4, see appendix D);
15. Severe neurological or psychiatric disease;
16. Significant hepatic dysfunction (serum bilirubin or transaminases ≥ 3 times the upper limit of normal (ULN)) unless related to hepatic involvement with MM.

    Note: Patients with Gilbert Syndrome are not excluded provided that direct bilirubin is ≤2 x ULN.
17. Significant renal dysfunction (creatinine clearance <30 ml/min after rehydration) Note: refer to Appendix F for creatinine clearance calculation;
18. Significant bone marrow suppression as evidenced by any of the below laboratory tests during screening:

    * Absolute neutrophil count ≤1.0 × 109/L;
    * Hemoglobin level ≤7.5 g/dL (≤4.65 mmol/L); transfusions are not allowed to reach this level
    * Platelet count ≤75 × 109/L in patients in whom <50% of bone marrow nucleated cells are plasma cells and platelet count ≤50 × 109/L in patients in whom ≥50% of bone marrow nucleated cells are plasma cells; transfusions are NOT allowed to reach this level
19. Concurrent severe and/or uncontrolled medical condition (e.g. uncontrolled diabetes, active systemic infection, uncontrolled hypertension, cancer, etc.) that is likely to interfere with the study procedures/results or which, in the opinion of the investigator, would constitute a hazard for participating in this study.
20. History of active malignancy during the past 5 years with the exception of basal carcinoma of the skin or stage 0 cervical carcinoma;
21. Any of the following:

    * Known active hepatitis A
    * Patient is seropositive for hepatitis B (defined by a positive test for hepatitis B surface antigen [HBsAg]). Patients with resolved infection (ie, patients who are positive for antibodies to hepatitis B core antigen [antiHBc] and/or antibodies to hepatitis B surface antigen [antiHBs]) must be screened using real-time polymerase chain reaction (PCR) measurement of hepatitis B virus (HBV) DNA levels. Those who are PCR positive will be excluded.

    EXCEPTION: Patients with serologic findings suggestive of HBV vaccination (antiHBs positivity as the only serologic marker) AND a known history of prior HBV vaccination, do not need to be tested for HBV DNA by PCR.

    o Known to be seropositive for hepatitis C (except in the setting of a sustained virologic response, defined as aviremia at least 12 weeks after completion of antiviral therapy).
22. Patient known to be HIV-positive;
23. Current participation in another clinical trial
24. Any psychological, familial, sociological and geographical condition potentially hampering compliance with the study protocol and follow-up schedule

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2019-10-31 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
CR or better | 5 years
  the proportion of patients who achieved CR or better

SECONDARY OUTCOMES:
Duration of Response | 5 years
  defined as time, in months, from initial response (PR or better) until the date of a disease progression event
Progression Free Survival | 5 years
  Progression Free Survival
Overall Response Rate | 5 years
  defined as the proportion of patients who will achieve PR or better, as per IMWG criteria
Overall Survival | 5 years
Safety (Adverse Events) | 5 years
  Adverse Events of the investigational combination treatment

CONTACTS AND LOCATIONS:
Locations (8):
- Greece (2):
  - University of Athens, Athens
  - Anticancer Hospital of Thessaloniki, Thessaloniki
- Italy (2):
  - University of Bologna, Bologna
  - Univerity of Turin, Torino
- Turkey (Türkiye) (4):
  - Ankara University, Ankara
  - Dokuz Eylul University, Balçova
  - Erciyes University, Kayseri
  - Marmara University, Pendik

IPD SHARING:
Plan to Share IPD: No